CLINICAL TRIAL: NCT04862416
Title: Safety, Tolerability and Plasmodium Falciparum Transmission-reducing Activity of R0.6C Vaccine Adjuvanted With Alhydrogel Alone or Combined With Matrix-M in Healthy Malaria-naïve Adults in the Netherlands
Brief Title: Safety and Efficacy of R0.6C Vaccine
Acronym: STOP-TRANS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Statens Serum Institut (Other); Novavax (Industry)
Responsible Party: Principal Investigator, Matthew McCall, dr. MBB McCall, Radboud University Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STOP-TRANS; 2021-000017-17 (EudraCT Number)
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Malaria; Malaria,Falciparum
Keywords: Transmission; Transmission blocking vaccine; Malaria; Plasmodium falciparum; R0.6C; Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: Study groups will be assigned sequentially to low and high doses of R0.6C Vaccine. Within each dose group, participants will be assigned randomly (1:1) to one of two adjuvant arms (either Alhydrogel alone or Alhydrogel + Matrix-M).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 1A 30μg R0.6C Alhydrogel (Experimental): 3 subjects will receive four vaccinations of 30 ug R0.6C Alhydrogel on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 1B 30μg R0.6C Alhydrogel + Matrix M1 (Experimental): 3 subjects will receive four vaccinations of 30 ug R0.6C Alhydrogel + Matrix M1 on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 2A 30μg R0.6C Alhydrogel (Experimental): 5 subjects will receive four vaccinations of 30 ug R0.6C Alhydrogel on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 2B 30μg R0.6C Alhydrogel + Matrix M1 (Experimental): 5 subjects will receive four vaccinations of 30 ug R0.6C Alhydrogel + Matrix M1 on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 3A 100μg R0.6C Alhydrogel (Experimental): 3 subjects will receive four vaccinations of 100 ug R0.6C Alhydrogel on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 3B 100μg R0.6C Alhydrogel + Matrix M1 (Experimental): 3 subjects will receive four vaccinations of 100 ug R0.6C Alhydrogel + Matrix M1 on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 4A 100μg R0.6C Alhydrogel (Experimental): 5 subjects will receive four vaccinations of 100 ug R0.6C Alhydrogel on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine
- 4B 100μg R0.6C Alhydrogel + Matrix M1 (Experimental): 5 subjects will receive four vaccinations of 100 ug R0.6C Alhydrogel + Matrix M1 on days 0, 28, 56 and 168.
  Interventions: Biological: R0.6C transmission blocking vaccine

INTERVENTIONS:
Biological: R0.6C transmission blocking vaccine — Vaccination with R0.6C transmission blocking vaccine. Volunteers will sequentially receive four administrations of R0.6C intramuscularly in the deltoid muscle on alternating sides on days 0, 28, 56 and 168.

SUMMARY:
This is a first-in-human phase I, open-label, single-site, dose escalation study to determine the safety, tolerability and Plasmodium falciparum transmission reducing activity of the R0.6C vaccine in two different adjuvant combinations.

DETAILED DESCRIPTION:
Thirty-two healthy adult volunteers will be recruited and divided over the study arms that will receive four vaccinations on days 0, 28, 56 and 168 with either 30μg or 100μg of R0.6C adjuvanted with Alhydrogel alone, or combined with Matrix-M1.

Three volunteers (Group 1A, n=3) will receive four vaccinations with the lower dose of 30μg R0.6C with Alhydrogel, and, in parallel, three volunteers (Group 1B, n=3) will receive four vaccinations with the lower dose of 30μg R0.6C with Alhydrogel and Matrix-M1. Volunteers will be closely monitored for adverse events for a period of minimally 14 days after the first vaccination. If safe, an additional 5 volunteers per adjuvant arm (groups 2A and 2B) will then receive four vaccinations with the lower dose (30μg R0.6C). If considered safe following a minimum of 14 days of follow-up after the first R0.6C administration of groups 2A and 2B, three volunteers per adjuvant arm (groups 3A and 3B) will start the vaccination regimen with the higher dose of 100μg R0.6C. Finally, a minimum of 14 days after administration of the first vaccination in groups 3A and 3B, if considered safe, an additional 5 volunteers per adjuvant arm (groups 4A and 4B) will initiate the vaccination regimen with the higher dose of 100μg R0.6C. There will be no placebo group. All volunteers will be followed up for adverse events until 84 days after the last immunisation. Total trial duration is approximately 8 months for each subject. Blood will be collected to assess functional Plasmodium falciparum transmission reducing activity (TRA) and transmission blocking activity (TBA) by standard membrane feeding assay (SMFA), as well as immunogenicity, at pre-specified time points after R0.6C vaccinations compared to pre-vaccination values.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must sign written informed consent to participate in the trial.
2. Subject is a male or non-pregnant and non-lactating female age ≥ 18 and ≤ 55 years and in good health.
3. Subject is able to understand planned study procedures and demonstrate comprehension of the protocol procedures and knowledge of study by passing a quiz (assessment of understanding).
4. In the opinion of the investigator, the subject can and will comply with the requirements of the protocol.
5. Subjects are available to attend all study visits and are reachable by phone throughout the entire study period from day -1 until day 224 (end of study).
6. The subject will remain within reasonable travelling distance from the study center from day -1 until day 7 after each R0.6C administration and agrees not to travel to a malaria-endemic area during the study period
7. Subject agrees to their general practitioner (GP) being informed about participation in the study and agrees to sign a form to request the release by their GP, and medical specialist when necessary, of any relevant medical information concerning possible contra-indications for participation in the study to the investigator(s).
8. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period according to current Sanquin guidelines.
9. Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause. All subjects of childbearing potential must agree to use continuous adequate contraception* until 2 months after completion of the study. Female subjects must agree not to breastfeed from 30 days prior to R0.6C administration until 2 months after completion of the study. Female subjects must have a negative pregnancy test at the inclusion visit.

Exclusion Criteria:

1. Acute or chronic disease at time of R0.6C administration, clinically significant pulmonary, cardiovascular, hepatic, renal, neurological or immunological functional abnormality, as determined by medical history, physical examination or laboratory screening tests:

   1. Acute disease is defined as the presence of a moderate or severe illness with or without fever. For subjects with an illness on the day of R0.6C administration, the vaccination may be postponed up to 7 days.
   2. Fever is defined as an oral, axillary or tympanic temperature ≥ 38.0°C.
   3. Any abnormal and clinically significant baseline laboratory screening tests of ALT, AST, creatinine, hemoglobin, platelet count or total white blood cell count, as defined in the protocol according to the FDA Toxicity Grading Scale for Healthy Adult and Adolescent Subjects Enrolled in Preventative Vaccine Clinical Trials (appendix 1).
2. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.
3. Chronic use of i) immunosuppressive drugs, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.
4. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or at inclusion.
5. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV).
6. Use of any other investigational or non-registered product (drug or vaccine) during the study period.
7. Known hypersensitivity to macrolides.
8. Participation in any other clinical study involving an investigational product in the 30 days prior to the start of the study or during the study period.
9. Receipt of any other vaccination within 30 days prior to the first R0.6C vaccination or planned vaccinations during the study period. Exceptions are made for vaccination against influenza and the novel coronavirus SARS-CoV2.
10. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study or CHMI.
11. Body weight > 115 kg
12. Being an employee or student of the department of Medical Microbiology of the Radboudumc at the time of screening, or a person otherwise related to the investigator.
13. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McCall, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Alkema M, Smit MJ, Marin-Mogollon C, Totte K, Teelen K, van Gemert GJ, van de Vegte-Bolmer M, Mordmuller BG, Reimer JM, Lovgren-Bengtsson KL, Sauerwein RW, Bousema T, Plieskatt J, Theisen M, Jore MM, McCall MBB. A Pfs48/45-based vaccine to block Plasmodium falciparum transmission: phase 1, open-label, clinical trial. BMC Med. 2024 Apr 23;22(1):170. doi: 10.1186/s12916-024-03379-y. PMID 38649867

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
Started | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5
Completed | 3 | 2 | 5 | 4 | 3 | 3 | 5 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1 | Total
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 22 [18 to 50] | 50 [19 to 53] | 23 [20 to 51] | 23 [23 to 44] | 27 [20 to 47] | 23 [20 to 23] | 21 [21 to 25] | 21 [18 to 49] | 23 [18 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 2 | 3 | 2 | 3 | 4 | 21
  Male | 2 | 1 | 1 | 3 | 0 | 1 | 2 | 1 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 2 | 3 | 5 | 4 | 3 | 3 | 5 | 5 | 30
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Brazilian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5 | 32
Weight (kg) [Median (Full Range); unit: kg] | 84.6 [72.0 to 90.0] | 69.2 [68.6 to 73.4] | 67.0 [57.0 to 77.4] | 74.0 [61.0 to 75.6] | 82.6 [64.0 to 89.0] | 68.0 [65.0 to 72.8] | 65.4 [57.8 to 80.5] | 63.8 [57.0 to 71.0] | 70.1 [57.0 to 90.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events and Grade 3 Adverse Events
Description: The number of serious adverse events and solicited and unsolicited grade 3 adverse events possibly, probably or definitely related to the vaccine in the period from first R0.6C administration up to 84 days after the last immunization.
Time Frame: From first immunization up to 84 days after the last immunization
Measure: Number; unit: adverse events
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5
adverse events
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Transmission Reducing Activity
Description: The functional transmission reducing activity in the standard membrane feeding assay of volunteer sera collected two weeks after the fourth R0.6C immunization (I4+14), compared to baseline (I1-1) within each of the four dose-adjuvant groups. The TRA was calculated by dividing the total number of oocysts in mosquitoes fed with I4+14 sera by total number of oocysts in mosquitoes fed with I1-1 sera.
Time Frame: 14 days after the fourth immunization
Measure: Median (Full Range); unit: % transmission reducing activity
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
Number analyzed (Participants) | 3 | 2 | 5 | 5 | 3 | 3 | 5 | 5
% transmission reducing activity | 17 [3 to 27] | -73 [-81 to -64] | -10 [-32 to 4] | -3 [-157 to 16] | 0 [-13 to 30] | -14 [-118 to 16] | 26 [-70 to 53] | 13 [-10 to 22]

3. Secondary Outcome: Number of Grade 1 and 2 Adverse Events
Description: The number of solicited and unsolicited grade 1 and 2 adverse events possibly, probably or definitely related to the vaccine in the period from first R0.6C administration up to 84 days after the last immunization.
Time Frame: From first immunization up to 84 days after the last immunization
Measure: Number; unit: adverse events
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
Number analyzed (Participants) | 3 | 3 | 5 | 5 | 3 | 3 | 5 | 5
adverse events | 11 | 18 | 33 | 61 | 17 | 51 | 32 | 69

4. Secondary Outcome: Transmission Reducing Activity
Description: The transmission reducing activity at other timepoint (I1+14, I2+14, I3+14, I3+111 [I4-1], and I4+84) compared to baseline (I1-1) in each of the four dose-adjuvant groups. The TRA was calculated by dividing the total number of oocysts in mosquitoes fed with I1+14, I2+14, I3+14, I3+111 [I4-1], and I4+84 sera by total number of oocysts in mosquitoes fed with I1-1 sera.
Time Frame: 14 days after immunization 1, 2 and 3. One day before immunization 4 and 84 days after immunization 4.
Population: TRA data were collected first for time points with highest antibody titres, if no significant TRA was detectable at these time points, TRA data was not collected for other timepoints.
Measure: Median (Full Range); unit: % transmission reducing activity
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
Number analyzed (Participants) | 3 | 2 | 5 | 5 | 3 | 3 | 5 | 5
% transmission reducing activity
  I3+14 | 3 [-6 to 10] | -80 [-99 to -61] | -3 [-19 to 27] | -9 [-16 to 22] | 15 [-21 to 28] | -42 [-63 to 30] | 16 [-20 to 43] | 9 [-69 to 51]
  I1+14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  I2+14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  I3+111 [I4-1]: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  I4+84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Anti-6C Antibody Quantities
Description: The anti-6C antibody quantity in volunteer sera collected two weeks after fourth R0.6C immunization (I4+14) and at other time points (I1+14, I2+14, I3+14, I3+111 [I4-1], and I4+84) compared to baseline (I1-1) in each of the four dose-adjuvant combinations, as determined by ELISA.
Time Frame: 14 days after each immunization. One day before immunization 4 and 84 days after immunization 4.
Population: One subject in group 2B withdrew consent 24 days after vaccination 4, therefore the I4+84 timepoint is only analyzed in 4 out of 5 subjects of group 2B.
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
Number analyzed (Participants) | 3 | 2 | 5 | 5 | 3 | 3 | 5 | 5
ug/mL
  I1-1 | 0.20 [0.10 to 0.30] | 0.24 [-0.18 to 0.66] | 0.21 [0.10 to 0.33] | 0.09 [0.05 to 0.12] | 0.25 [0.08 to 0.43] | 0.12 [0.09 to 0.14] | 0.11 [0.01 to 0.21] | 0.09 [0.02 to 0.16]
  I1+14 | 0.23 [0.14 to 0.31] | 0.21 [-0.21 to 0.64] | 0.27 [0.00 to 0.54] | 0.11 [0.05 to 0.17] | 0.20 [0.05 to 0.36] | 0.18 [0.07 to 0.28] | 0.11 [-0.01 to 0.22] | 0.21 [0.14 to 0.28]
  I2+14 | 0.33 [0.17 to 0.48] | 1.62 [0.20 to 3.03] | 0.42 [0.24 to 0.59] | 4.42 [-13.84 to 22.69] | 0.78 [0.11 to 1.45] | 3.26 [2.75 to 3.78] | 0.27 [0.00 to 0.54] | 3.52 [-1.13 to 8.18]
  I3+14 | 0.87 [-0.91 to 2.64] | 2.57 [1.81 to 3.33] | 1.20 [-0.98 to 3.38] | 4.39 [-6.13 to 14.91] | 1.67 [0.80 to 2.54] | 5.64 [4.12 to 7.17] | 0.59 [-0.14 to 1.33] | 5.56 [-0.42 to 11.53]
  I4-1 | 0.38 [0.30 to 0.46] | 0.58 [-0.29 to 1.45] | 0.42 [0.25 to 0.59] | 0.79 [-0.21 to 1.79] | 0.46 [0.32 to 0.59] | 0.86 [0.63 to 1.10] | 0.24 [0.01 to 0.47] | 0.73 [0.25 to 1.22]
  I4+14 | 1.61 [-1.43 to 4.65] | 5.22 [1.22 to 9.22] | 2.31 [1.56 to 3.07] | 4.13 [-3.52 to 11.78] | 2.40 [-1.34 to 6.14] | 7.57 [3.46 to 11.68] | 1.73 [-0.65 to 4.11] | 5.75 [0.26 to 11.24]
  I4+84: number analyzed (Participants) | 3 | 2 | 5 | 4 | 3 | 3 | 5 | 5
  I4+84 | 0.76 [0.00 to 1.51] | 1.96 [0.22 to 3.71] | 0.85 [0.57 to 1.13] | 1.69 [-2.09 to 5.48] | 1.04 [0.53 to 1.55] | 1.74 [0.96 to 2.51] | 0.58 [-0.10 to 1.26] | 2.10 [0.56 to 3.64]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from baseline until 84 days after the fourth vaccination (252 days).
Arm/Group | 1A 30μg R0.6C Alhydrogel | 1B 30μg R0.6C Alhydrogel + Matrix M1 | 2A 30μg R0.6C Alhydrogel | 2B 30μg R0.6C Alhydrogel + Matrix M1 | 3A 100μg R0.6C Alhydrogel | 3B 100μg R0.6C Alhydrogel + Matrix M1 | 4A 100μg R0.6C Alhydrogel | 4B 100μg R0.6C Alhydrogel + Matrix M1
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/5 | 0/3 | 0/3 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/5 | 0/3 | 0/3 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 5/5 | 3/3 | 3/3 | 5/5 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A 30μg R0.6C Alhydrogel (N=3) | 1B 30μg R0.6C Alhydrogel + Matrix M1 (N=3) | 2A 30μg R0.6C Alhydrogel (N=5) | 2B 30μg R0.6C Alhydrogel + Matrix M1 (N=5) | 3A 100μg R0.6C Alhydrogel (N=3) | 3B 100μg R0.6C Alhydrogel + Matrix M1 (N=3) | 4A 100μg R0.6C Alhydrogel (N=5) | 4B 100μg R0.6C Alhydrogel + Matrix M1 (N=5)
Pain at injection site (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (3) | 5 (14) | 4 (13) | 3 (9) | 3 (12) | 5 (20) | 5 (20)
Induration at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 4 (5) | 1 (3) | 3 (6) | 0 (0) | 3 (8)
Itching at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 4 (7) | 1 (1) | 3 (6) | 0 (0) | 5 (12)
Erythema at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 5 (12) | 1 (2) | 3 (7) | 0 (0) | 4 (10)
Swelling at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 1 (1) | 3 (5)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (6) | 2 (4) | 1 (1) | 1 (2) | 4 (6) | 2 (5)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (2) | 2 (5) | 4 (34) | 4 (23) | 2 (4) | 2 (15) | 1 (6) | 2 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3) | 1 (2) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tenderness at injection site (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Drowsiness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated leukocytes (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tired sensation vaccinated upper arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (2) | 2 (4) | 2 (3)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushes (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain between shoulder blades (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in armpit (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Common cold (Infections and infestations) | 1 (2) | 2 (2) | 4 (8) | 4 (9) | 2 (4) | 2 (2) | 2 (2) | 3 (9)
Herpes simplex infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 3 (3) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma after venipuncture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Spotting (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichomonas infection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hay fever (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otalgia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thoracic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cut wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04862416/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT04862416/SAP_001.pdf
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04862416/ICF_002.pdf